CLINICAL TRIAL: NCT00222378
Title: Prevalence of Cytomegalovirus, Epstein Barr Virus and Human Herpes 6 Virus DNA in Intestinal Mucosa of Patients With Inflammatory Bowel Disease
Brief Title: Prevalence of Cytomegalovirus, Epstein Barr Virus and Human Herpes 6 Virus in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Paul Feldman, Assistant Professor, University of Miami
Other Study IDs: 20043510; Protocol VAL094; WIRB® Protocol #20050561 (Other: WIRB)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-05

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease; ulcerative colitis; cytomegalovirus; Epstein Bar Virus; Human Herpes virus 6
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be discarded upon study completion
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An increase prevalence of CMV, EBV and or HHV-6 in diseased tissue of inflammatory bowel disease would suggest a role for these viruses in the etiology and/or exacerbation of IBD, whereas their absence would preclude such association.

DETAILED DESCRIPTION:
The protocol is designed to evaluate the following objectives:

1. The prevalence of cytomegalovirus, Epstein Barr virus and human herpes 6 virus DNA in inflamed intestinal mucosa of patients with Crohn's colitis and ulcerative colitis compared to their prevalence in healthy intestinal mucosa of patients not affected by these conditions;
2. To evaluate the prevalence of cytomegalovirus, Epstein Barr virus and human herpes 6 virus DNA in the intestinal mucosa of patients with Crohn's colitis and ulcerative colitis compared to that in inflamed mucosa caused by other conditions (non specific colitis);
3. To compare the prevalence of cytomegalovirus, Epstein Barr virus and human herpes 6 virus DNA in inflamed and healthy tissue in the same patients with Crohn's colitis and ulcerative colitis;
4. To determine whether the presence of cytomegalovirus, Epstein Barr virus and human herpes 6 virus DNA detected by nPCR correlates with immunohistochemical detection of viral protein in colonic tissue.
5. To determine whether the relative viral quantity of CMV, EBV or HHV-6 is related to severity of disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Documented, signed and dated informed consent to participate in this trial prior to any study related procedures being performed.
* Participants, male or female, aged 18-70, identified as having Crohn's colitis, UC and patients undergoing biopsy for other inflammatory disorders (non specific colitis) and for suspected intestinal malignancy.

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) infection
* Post organ transplant patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease (ulcerative colitis and Crohn's Colitis), Other inflammatory conditions of the colon
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2005-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of Cytomegalovirus and Epstein Barr Virus in Patients with Mild to Moderate Inflammatory Bowel Disease compared to patients without inflammatory bowel disease | 0
Prevalence of Cytomegalovirus and Epstein Barr Virus in inflamed colonic tissue versus non inflamed tissues from Patients with Mild to Moderate Inflammatory. | 0
Prevalence of Cytomegalovirus and Epstein Barr Virus in inflamed colonic tissue from patient with mild to moderate IBD as compared to inflamed mucosa from patients with other inflammatory diseases of the colon | 0

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Raskin, M.D., Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

REFERENCES:
- [Background] Wakefield AJ, Fox JD, Sawyerr AM, Taylor JE, Sweenie CH, Smith M, Emery VC, Hudson M, Tedder RS, Pounder RE. Detection of herpesvirus DNA in the large intestine of patients with ulcerative colitis and Crohn's disease using the nested polymerase chain reaction. J Med Virol. 1992 Nov;38(3):183-90. doi: 10.1002/jmv.1890380306. PMID 1287131
- [Background] Berk T, Gordon SJ, Choi HY, Cooper HS. Cytomegalovirus infection of the colon: a possible role in exacerbations of inflammatory bowel disease. Am J Gastroenterol. 1985 May;80(5):355-60. PMID 2859801
- [Background] el-Serag HB, Zwas FR, Cirillo NW, Eisen RN. Fulminant herpes colitis in a patient with Crohn's disease. J Clin Gastroenterol. 1996 Apr;22(3):220-3. doi: 10.1097/00004836-199604000-00015. PMID 8724263
- [Background] Caserta L, Riegler G. Cytomegalovirus and herpes simplex virus antibodies in patients with idiopathic ulcerative colitis. Am J Gastroenterol. 2001 Oct;96(10):3036-7. doi: 10.1111/j.1572-0241.2001.04690.x. No abstract available. PMID 11693350
- [Background] Riegler G, Piscitelli A, Di Simone A, Esposito C, Sodano G, Tarro G. [Cytomegalovirus and herpes simplex virus antibodies in patients with idiopathic ulcerative rectocolitis]. Minerva Med. 1990 Dec;81(12):861-4. Italian. PMID 2177863
- [Background] Cooper HS, Raffensperger EC, Jonas L, Fitts WT Jr. Cytomegalovirus inclusions in patients with ulcerative colitis and toxic dilation requiring colonic resection. Gastroenterology. 1977 Jun;72(6):1253-6. PMID 192627
- [Background] Sidi S, Graham JH, Razvi SA, Banks PA. Cytomegalovirus infection of the colon associated with ulcerative colitis. Arch Surg. 1979 Jul;114(7):857-9. doi: 10.1001/archsurg.1979.01370310099019. PMID 222233
- [Background] Cottone M, Pietrosi G, Martorana G, Casa A, Pecoraro G, Oliva L, Orlando A, Rosselli M, Rizzo A, Pagliaro L. Prevalence of cytomegalovirus infection in severe refractory ulcerative and Crohn's colitis. Am J Gastroenterol. 2001 Mar;96(3):773-5. doi: 10.1111/j.1572-0241.2001.03620.x. PMID 11280549
- [Background] Adani GL, Avital I, Ferraresso C, Aoki T. CMV infection in severe refractory ulcerative and Crohn's colitis. Am J Gastroenterol. 2001 Dec;96(12):3464-5. doi: 10.1111/j.1572-0241.2001.05360.x. No abstract available. PMID 11774988
- [Background] Wada Y, Matsui T, Matake H, Sakurai T, Yamamoto J, Kikuchi Y, Yorioka M, Tsuda S, Yao T, Yao S, Haraoka S, Iwashita A. Intractable ulcerative colitis caused by cytomegalovirus infection: a prospective study on prevalence, diagnosis, and treatment. Dis Colon Rectum. 2003 Oct;46(10 Suppl):S59-65. doi: 10.1097/01.DCR.0000087486.21981.C6. PMID 14530660
- [Background] Kambham N, Vij R, Cartwright CA, Longacre T. Cytomegalovirus infection in steroid-refractory ulcerative colitis: a case-control study. Am J Surg Pathol. 2004 Mar;28(3):365-73. doi: 10.1097/00000478-200403000-00009. PMID 15104299
- [Background] Probert CS, Hearing SD, Schreiber S, Kuhbacher T, Ghosh S, Arnott ID, Forbes A. Infliximab in moderately severe glucocorticoid resistant ulcerative colitis: a randomised controlled trial. Gut. 2003 Jul;52(7):998-1002. doi: 10.1136/gut.52.7.998. PMID 12801957
- [Background] Bertalot G, Villanacci V, Gramegna M, Orvieto E, Negrini R, Saleri A, Terraroli C, Ravelli P, Cestari R, Viale G. Evidence of Epstein-Barr virus infection in ulcerative colitis. Dig Liver Dis. 2001 Oct;33(7):551-8. doi: 10.1016/s1590-8658(01)80106-7. PMID 11816543
- [Background] Spieker T, Herbst H. Distribution and phenotype of Epstein-Barr virus-infected cells in inflammatory bowel disease. Am J Pathol. 2000 Jul;157(1):51-7. doi: 10.1016/S0002-9440(10)64516-6. PMID 10880375
- [Background] Yanai H, Shimizu N, Nagasaki S, Mitani N, Okita K. Epstein-Barr virus infection of the colon with inflammatory bowel disease. Am J Gastroenterol. 1999 Jun;94(6):1582-6. doi: 10.1111/j.1572-0241.1999.01148.x. PMID 10364028